CLINICAL TRIAL: NCT06841965
Title: Th Efficacy and Safety of Intravenous Thrombolysis in Acute Ischemic Stroke with Cancer
Brief Title: Intravenous Thrombolysis in Acute Ischemic Stroke with Active Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICE
Record Dates: First submitted 2025-01-20; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous thrombolysis (alteplase and other guideline-recommended thrombolytic agents)) (Experimental): Patients will receive standard dose intravenous alteplase (0.9 mg/kg, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)，intravenous Tenecteplase(0.25mg/kg，administered as a single intravenous bolus injection over 5 - 10 seconds，with a maximum dose of 25 mg), intravenous reteplase (a bolus of 18 mg followed by a second bolus of 18 mg after 30 minutes) and intravenous prourokinase (rhPro-UK) (15 mg bolus followed by a 20 mg infusion over 30 minutes).
  Interventions: Drug: Intravenous thrombolysis
- Standard therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Intravenous thrombolysis — Patients will receive standard dose intravenous alteplase (0.9 mg/kg, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)，intravenous Tenecteplase(0.25mg/kg，administered as a single intravenous bolus injection over 5 - 10 seconds，with a maximum dose of 25 mg), intravenous reteplase (a bolus of 18 mg followed by a second bolus of 18 mg after 30 minutes) and intravenous prourokinase (rhPro-UK) (15 mg bolus followed by a 20 mg infusion over 30 minutes).
  Arms: Intravenous thrombolysis (alteplase and other guideline-recommended thrombolytic agents))

SUMMARY:
The primary hypothesis being tested in this trial is that ischemic stroke patients with active cancer will have improved clinical outcomes when given intravenous thrombolysis compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical signs of acute ischemic stroke within 24 hours of onset or awakening with stroke (if within 24 hours from the midpoint of sleep). Patients with AIS within 4.5-24 hours of onset must meet the IVT inclusion criteria specified in the guideline
2. Patients with active cancer (Active cancer was defined as cancer diagnosed within the previous 6 months; recurrent, regionally advanced or metastatic cancer, or cancer for which treatment had been administered within 6 months, or haematological cancer without complete remission.)
3. Patients ≥ 18 years old
4. Informed consent has been obtained depending on local ethics requirements.

Exclusion Criteria:

(1) Intended to proceed to endovascular treatment; (2) Pre-stroke mRS score > 2 (3) Contraindications for IVT：

1. Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, epidural hematoma, etc.)
2. Previous history of intracranial hemorrhage
3. Severe head trauma or stroke history within the last 3 months
4. Intracranial tumors, giant intracranial aneurysms
5. Intracranial or spinal surgery within the recent 3 months
6. Major surgical procedures within the last 2 weeks
7. Gastrointestinal or urinary tract bleeding within the last 3 weeks
8. Active visceral bleeding
9. Aortic arch dissection
10. Arterial puncture in a site within the last 1 week that is not easy to compress and stop bleeding
11. Elevated blood pressure: Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg
12. Acute bleeding tendency, including platelet count < 100 × 10⁹/L or other conditions
13. Received low-molecular-weight heparin treatment within 24 hours
14. Oral anticoagulants (warfarin) with INR > 1.7 or PT > 15 s; Receiving heparin treatment with aPTT above the upper limit of the normal range within the last 24 hours of onset, Receiving thrombin inhibitors and factor Xa inhibitors within the last 48 hours of onset.
15. Blood sugar < 2.8 or > 22.22 mmol/L
16. Head CT or MRI indicates large-area infarction (infarction area ≥ 1/3 of the middle cerebral artery supply area) (4) The judgment is left to the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Independent recovery assessed by ratio of modefied Rankin Scale (mRS) score of 0-2 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
Excellent recovery assessed by the ratio of modified Rankin Scale (mRS) score of 0-1 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
recovery assessed by modefied Rankin Scale (mRS) score | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
3-month mortality | 90 ± 7 days
  Hospitalization records or follow-up results
Presence of parenchymal hemorrhage (PH) evaluated by CT or MRI | at day 1
  the presence of PH is defined according the standard from ECASS-2 study
Presence of symptomatic intracerebral hemorrhage (sICH) evaluated by CT or MRI | at day 1
  the presence of sICH is defined according the standard from ECASS-2 study
Presence of hemorrhagic transformation evaluated by CT or MRI | at day 1
  Presence of hemorrhagic transformation is defined according the standard from ECASS-2 study

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, PhD, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No
Protecting the privacy of participants is a priority, and sharing IPD could potentially compromise this.